CLINICAL TRIAL: NCT02730975
Title: Pharmacokinetic Food-effect Study of Abiraterone Acetate (A.A) in Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: Pharmacokinetic Food-effect Study of Abiraterone Acetate (AA) in Castration Resistant Prostate Cancer
Acronym: ABIFOOD01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABIFOOD01; 2012-003226-25 (EudraCT Number)
Record Dates: First submitted 2015-09-15; First posted 2016-04-07 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Prostate Cancer
Keywords: pharmacokinetics; food-effect; fat diet; abiraterone acetate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AA Reduced dose-normal diet (A) (Experimental): Abiraterone acetate at reduced dose of 250 mg po daily in cycles of 28 days administered with a standard breakfast
  Interventions: Drug: AA Reduced dose-normal diet (A)
- AA reduced dose-fat diet (B) (Experimental): Abiraterone acetate at reduced dose of 250 mg po daily in cycles of 28 days administered with a fat breakfast
  Interventions: Drug: AA reduced dose-fat diet (B)
- AA normal dose-fasting conditions (C) (Active Comparator): Abiraterone acetate at approved dose of 1000 mg po daily in cycles of 28 days administered in fasting conditions
  Interventions: Drug: AA normal dose-fasting conditions (C)

INTERVENTIONS:
Drug: AA Reduced dose-normal diet (A) — Cycles of 28 days length of AA at reduced doses (250 mg) administered with a pre-defined normal diet, described with specific caloric and fat content.
  Other Names: Abiraterone acetate 250 mg normal diet
  Arms: AA Reduced dose-normal diet (A)
Drug: AA reduced dose-fat diet (B) — Cycles of 28 days length of AA at reduced doses (250 mg) administered with a pre-defined fat diet, described with specific caloric and fat content.
  Other Names: Abiraterone acetate 250 mg fat- diet
  Arms: AA reduced dose-fat diet (B)
Drug: AA normal dose-fasting conditions (C) — Cycles of 28 days length of AA at approved doses (1000 mg) administered in fasting conditions.
  Other Names: Abiraterone acetate 1000 mg fasting conditions
  Arms: AA normal dose-fasting conditions (C)

SUMMARY:
ABIFOOD study is a randomized open-labelled, phase I study to evaluate food effect in the pharmacokinetic parameters of abiraterone acetate (AA) at reduced doses, versus AA in fasting conditions at conventional doses, in castration resistant prostate cancer (mCRPC) patients who have progressed to docetaxel.

DETAILED DESCRIPTION:
Abiraterone acetate (AA) has been approved for the treatment of mCRPC after docetaxel progression at doses of 1.000 mg per day taken in fasting conditions. However, it has been described both the significant food-effect on bioavailability up to 5 to 10 times folder increase depending on the fat content of the diet. These data come from the analysis of a small number of patients in phase I studies conducted in the early stages of drug development and some exploratory study in healthy subjects. There is not prospective randomized study that has analyzed the real impact of the normal diet in the bioavailability of the drug (not a fatty diet like has been used in initial studies).

Given the particular epidemiology of mCRPC (relatively frequent pathology), and taking into account recent data which indicates positive results of AA treatment in patients who had not previously received chemotherapy, a significant use of this drug is anticipated in the uro-oncology community in the coming years.

The precise definition of dose according to the food-effect on bioavailability may be critical not only from a purely medical perspective and / or pharmacological but even for its socioeconomic impact in our health system.

The hypothesis for this study is to prove that AA administered in reduced doses with standard diet presents a suitable pharmacokinetic profile which would achieve therapeutic levels in blood, so that regimens lower than currently approved in association with food can be used in future studies on efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed prostate adenocarcinoma without neuroendocrine differentiation or with no small cell histology.
* At least one, but no more than two regimens of cytotoxic chemotherapy for metastatic castration-resistant prostate cancer. At least one regimen must have contained docetaxel.
* Men 18 years old or more.
* Criteria for progression according to the recommendations of the Prostate Cancer Working Group.
* Androgen deprivation present with testosterone levels <50 ng / dl or <2.0 nmol / l).
* ECOG (Eastern Cooperative Oncology Group) performance status <2.
* Adequate organ function
* Accept the use of barrier methods of contraception throughout the study
* Signature of informed consent to participate in the study consent.

Exclusion Criteria:

* Inability or unwillingness to swallow tablets.
* Known brain metastases
* Significant chronic gastrointestinal disorder with diarrhea as the main symptom (Crohn's disease, ulcerative colitis, malabsorption, or grade ≥ 2 diarrhea of any etiology at baseline).
* Local prostate surgery or intervention within 30 days prior to the first dose. Further, any clinically relevant sequel to surgery should be resolved before the 1st of cycle 1.
* Radiotherapy, chemotherapy or immunotherapy within 30 days before or single fraction of palliative radiotherapy within 14 days prior to the administration of the day 1of Cycle 1.
* Patients with uncontrolled hypertension, clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, heart failure Class III or IV of the New York Heart Association or cardiac ejection fraction <50%, active or symptomatic viral hepatitis, chronic liver failure, clinically significant adrenal or pituitary dysfunction. (Patients with hypertension controlled with drugs are allowed)
* Any acute toxicity due to chemotherapy and / or prior radiotherapy has not been resolved to ≤ grade 1 NCI CTCAE (version 4). Alopecia and grade 2 peripheral neuropathy induced by chemotherapy are allowed.
* Previous treatment with abiraterone acetate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-05-12 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) | 1, 2, 3, 4, 5, 6, 8, 12, y 24 hours post dose in day 1 of cycle 1 (28 days long) , day 10-14 of cycle 1 and day 1 of cycle 5(28 days long)
  Area under curve at time t and infinite, compared with abiraterone acetate administered a standard dose fasting in the times specified: 1, 2, 3, 4, 5, 6, 8, 12, y 24 hours post dose
Peak Plasma Concentration (Cmax) | 1, 2, 3, 4, 5, 6, 8, 12, y 24 hours post dose in day 1 of cycle 1 (28 days long) , day 10-14 of cycle 1 and day 1 of cycle 5(28 days long)
  Peak Plasma Concentration (Cmax) of acetate administered at low doses with meals, compared with abiraterone acetate administered a standard dose fasting in the times specified: 1, 2, 3, 4, 5, 6, 8, 12, y 24 hours post dose
Time to reach peak plasma concentration (Tmax) | 1, 2, 3, 4, 5, 6, 8, 12, y 24 hours post dose in day 1 of cycle 1 (28 days long) , day 10-14 of cycle 1 and day 1 of cycle 5(28 days long)
  Time to reach peak plasma concentration (Tmax) of acetate administered at low doses with meals, compared with abiraterone acetate administered a standard dose fasting in the times specified: 1, 2, 3, 4, 5, 6, 8, 12, y 24 hours post dose

SECONDARY OUTCOMES:
PSA (Prostate Specific Antigen) levels | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Basal PSA levels and monitoring until disease progression
Response rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Response rate according to RECIST 1.1
Pain intensity | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Pain intensity measured by the Brief Pain Inventory-Short Form scale (BPI-SF)
Use of analgesics | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Type of analgesics used for pain treatment.
Total daily dose of analgesics | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Total daily dose of analgesics will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Durán Martínez, MD-PhD, Study Director — Hospital Universitario Virgen del Rocío, Seville, Spain; Clara Rosso Fernández, MD-PhD, Principal Investigator — Hospital Universitario Virgen del Rocío, Seville, Spain
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided